CLINICAL TRIAL: NCT06247657
Title: A Phase I, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of BL0006 as a Single Agent in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study to Assess the Safety and Tolerability of BL0006 for Patients With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Best-Link Bioscience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL0006-101
Record Dates: First submitted 2024-01-10; First posted 2024-02-08 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL0006 (Experimental): Patients will be administered BL0006 via intravenous infusion at the corresponding dose level on days 1 and 8 of a 21-days treatment cycle.
  Interventions: Drug: BL0006

INTERVENTIONS:
Drug: BL0006 — Patients will be administered BL0006 via intravenous infusion at the corresponding dose level on days 1 and 8 of a 21-days treatment cycle.

SUMMARY:
This is the first in human study of BL0006, and the primary objective is to evaluate the safety and tolerability of BL0006 as a single agent in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study consists of two parts: dose-escalation stage and dose-expansion stage.

The dose-escalation stage is designed to determine the maximum tolerated dose (MTD) and select recommended Phase 2 dose (RP2D) of BL0006 monotherapy. The dose-expansion stage will be conducted with selected doses to further evaluate the preliminary anti-tumor activity, safety and tolerability.

A total of approximately 19~66 patients will be enrolled in the study.

Approximately 13-30 patients will be enrolled into dose-escalation of BL0006 . A total of 6~36 patients each with advanced solid tumor will be evaluated in dose-expansion of BL0006.

Patients will continue to receive BL0006 as long as they are benefiting from treatment in the investigator's opinion and do not meet any other discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study, be able to understand the requirements of a clinical study, and sign informed consent form.
2. Aged ≥ 18 years, male and female.
3. The dose-escalation stage: patients with histologically or cytologically confirmed, unresectable or metastatic advanced solid tumors that have failed despite standard therapy, for whom no standard therapy exists, or who have refused standard therapy.
4. The dose-expansion stage: patients with histologically or cytologically confirmed, unresectable or metastatic hepatocellular carcinoma (HCC) who are not suitable for surgery and local treatment, and who have failed despite standard therapy, or who have refused standard therapy. And other potential tumors (selection based on the results of BL0006-101 Study dose-escalation stage) that have failed despite standard therapy, for whom no standard therapy exists, or who have refused standard therapy.
5. Patients with at least one measurable lesion per RECIST (v1.1) (applicable to the dose-expansion stage only).
6. Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1 at screening.
7. Life expectancy period ≥ 12 weeks.
8. A male patient must agree to use adequate contraception from screening through at least 6 months after the last dose of investigational product BL0006.
9. Women of childbearing potential must have a negative pregnancy test prior to the dosing administration, and agree to use adequate contraception from screening through at least 6 months after the last dose of investigational product BL0006. A female participant of non-childbearing potential will have had at least 12 continuous months of natural (spontaneous) amenorrhoea, follicle stimulating hormone (FSH) level > 40 mIU/mL at screening, and an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms); or have had surgical bilateral oophorectomy, hysterectomy or bilateral tubal ligation beyond 6 weeks prior to screening.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) metastases or carcinomatous meningitis.
2. Patients who have a history of another primary malignancy (with the exception of subjects with cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of uterine cervix). A patient who has had no evidence of disease from another primary cancer for 5 or more years is allowed to participate in the study.
3. Patients whose pericardial effusion, pleural effusion or ascites remain uncontrollable after intervention.
4. Patients with a history of allogeneic transplantation of organs, bone marrow or stem cell. Patients with a history of hepatic encephalopathy.
5. Patients with Gilbert's syndrome disease.
6. Patients with homozygous for UGT1A1*28 or UGT1A1*6.
7. Patients who have impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   New York Heart Association class III-IV for cardiac insufficiency or left ventricular ejection fraction < 50%.

   Patients with poorly controlled arrhythmia: QTc interval > 480 ms calculated by Fridericia's formula, or congenital syndrome of prolonged QT interval.

   Any of the following within 6 months prior to the screening: myocardial infarction, severe or unstable angina, congestive heart failure, cerebrovascular accident (including transient ischemic attack), symptomatic pulmonary embolism or other clinically significant thromboembolic disease, or coronary artery bypass graft.

   Clinically significant resting bradycardia. Patients with other clinically significant cardiovascular disease who were assessed as unsuitable for this study by the investigator.
8. Patients with active chronic inflammatory bowel disease at screening (such as Ulcerative Colitis, Crohn's disease), ≥ grade 2 anorexia, nausea, vomiting or signs of intestinal obstruction. Or patients with a history of intestinal obstruction, gastrointestinal perforation, or clinically significant gastrointestinal bleeding within the 6 months prior to screening.
9. Known history of clinically significant active Chronic Obstructive Pulmonary Disease (COPD), or other moderate-to-severe chronic respiratory illness present within 6 months.
10. Patients who have a known diagnosis of Human Immunodeficiency Virus (HIV) infection.
11. Patients with active hepatitis C or chronic hepatitis B at screening ("active hepatitis" defined as HCV RNA level ≥ 200 IU/mL for hepatitis C or HBV DNA level ≥ 2000 IU/mL for hepatitis B at screening). In addition, eligible hepatitis B or hepatitis C patients must agree to antiviral treatment according to the treatment guidelines.
12. Active infections requiring antibiotic intravenous therapy within 4 weeks prior to screening.
13. Patients with any other medical conditions that, in the opinion of the Investigator, could affect the patient's participation in the study such as:

    Disease management may be jeopardized by treatment with this study treatment. Uncontrolled diabetes mellitus, HbA1c ≥ 8%. Moderate or severe hepatic impairment, i.e., Child-Pugh class B or C.
14. Those who received blood transfusion, albumin, recombinant human thrombopoietin, or colony-stimulating factor therapy within 2 weeks prior to screening.
15. Patients who have not sufficient baseline organ function and whose laboratory data meet the following criteria at enrollment:

    Absolute Neutrophil Count (ANC) < 1.5×109/L. Serum albumin < 30 g/L. Total bilirubin > 1.5×ULN. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3×ULN without liver metastases or primary liver cancer. AST or ALT > 5×ULN if the patient has documented primary liver cancer or liver metastases.

    Hemoglobin < 90 g/L. Platelets < 100×109 /L. Creatinine clearance < 50 mL/min.
16. Those who are known to be allergic to the active ingredient or excipients of the investigational product BL0006, or who have a predisposition to allergy.
17. Patients with a history of an anaphylactic reaction to irinotecan, irinotecan liposome, sacituzumab govitecan-hziy or other topoisomerase I inhibitors, or ≥ Grade 3 hematology or gastrointestinal toxicity prior to irinotecan, irinotecan liposome, sacituzumab govitecan-hziy or other topoisomerase I inhibitors.
18. Use of UGT1A1 inhibitors or inducers within 5 half-lives at the time of investigational product BL0006 administration, or planned use of UGT1A1 inhibitors or inducers within 2 weeks prior to administration of BL0006 (whichever is shorter), or are expected to continue such therapy during the study.
19. Anti-tumor therapy within 5 half-lives at the time of investigational product BL0006 administration, or anti-tumor therapy within 4 weeks prior to administration of BL0006 (whichever is shorter), therapy including chemotherapy, biologic therapy, immunotherapy, radiotherapy (palliative radiotherapy for local pain control is excluded and the radiotherapy area do not include the proposed target lesion) and so on, or all relevant toxic reactions (except alopecia) have not been recovered.
20. Patients who are taking anticoagulant therapy (prophylactic use of low-dose aspirin or low molecular weight heparin is allowed).
21. Those who are expected to require systemic corticosteroids within 4 weeks prior to administration of BL0006 (low doses of corticosteroids are excluded, such as ≤ 10 mg prednisone daily or equivalent).
22. Those who have received live or attenuated vaccines (e.g., measles, mumps, rubella, varicella, yellow fever, rabies, BCG, typhoid vaccine, etc.) within 4 weeks before screening, or any covid-19 vaccine within 2 weeks before screening.
23. Those who underwent major surgery within 4 weeks before screening, or plan to undergo major surgery during the study.
24. Those who are participating in other clinical studies, or have participated in any other interventional clinical studies within 4 weeks before screening.
25. Pregnant or lactating women.
26. Patients who are judged disqualified to join clinical studies by investigator due to any causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD) | Throughout the study for approximately 2 years
  Based on the incidence of Dose-Limiting Toxicity (DLT) of BL0006 in patients with advanced solid tumors, MTD is determined.
Recommended Phase II Dose(RP2D) | Throughout the study for approximately 2 years
  RP2D will be evaluated according to all the available safety, PK and efficacy data.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | Cycle 1 day 1 to Cycle 2 day 2（each cycle is 21 days）
  Area under the plasma concentration time curve
Half life (t1/2) | Cycle 1 day 1 to Cycle 2 day 2（each cycle is 21 days）
  The elimination half-life time
Disease Control Rate(DCR) | Throughout the study for approximately 2 years
  DCR is defined as the proportion of subjects who achieve a Complete Response (CR) 、Partial Response (PR) or Stable Disease (SD) as assessed by RECIST v1.1
Objective response rate(ORR) | Throughout the study for approximately 2 years
  ORR is defined as the proportion of patients with the best responses of Complete Response (CR) and Partial Response (PR) observed after study treatment.
Progression-Free Survival (PFS) | Throughout the study for approximately 2 years
  PFS was defined as the the time from the start date of study treatment to the first documented disease progression or death due to any cause, whichever occurs first.
Duration of overall response (DOR) | Throughout the study for approximately 2 years
  DOR is defined as the time from the first documented CR or PR per RECIST v1.1 to disease recurrence or disease progression (PD) whichever occurs first.
One-year Overall Survival rate (OS 12) | Throughout the study for approximately 2 years
  OS 12 is defined as the proportion of patients alive at one year after the start date of study treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Hospital of Jilin University, Changchun, Jilin
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality